CLINICAL TRIAL: NCT03250793
Title: Physiologic Pilot Study: Work of Breathing Description in Neonates With Congenital Diaphragmatic Hernia in Post-surgical Period Alternatively in Conventional Ventilation (Pressure Controlled) and in NAVA (Neurally Adjusted Ventilatory Assist) Ventilation.
Brief Title: Work of Breathing Description in Neonates With Congenital Diaphragmatic Hernia in NAVA and in Conventional Ventilation.
Acronym: NAVA-DIAPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL17_0429; 2017-A02270-53 (Other: ID-RCB)
Record Dates: First submitted 2017-08-03; First posted 2017-08-16 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Hernia, DIaphragmatic, Congenital
Keywords: Hernia, DIaphragmatic, Congenital; Respiration, Artificial; physiologic pilot study; NAVA; Neurally Adjusted Ventilatory Assist; esophageal transducer; Work of Breathing
MeSH Terms: conditions — Hernia, Diaphragmatic; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neonate with congenital diaphragmatic hernia (Experimental): Neonates with congenital diaphragmatic hernia in post-surgical period under mechanical ventilation during weaning of mechanical ventilation
  Interventions: Device: Physiologic study measuring work of breathing which can be estimated by the esophageal and trans-diaphragmatic pressure-time product obtained by an esophageal transducer

INTERVENTIONS:
Device: Physiologic study measuring work of breathing which can be estimated by the esophageal and trans-diaphragmatic pressure-time product obtained by an esophageal transducer — While the patient is under respiratory assistance on the SERVO-I respirator, he will be included in the study and one esophageal transducer of 2,3 mm of diameter will be inserted through the mouth / nose in addition to NAVA's naso / Oro-Gastric tube( Edi Catheter, 6Fr, 49 cm, PHT free 5 pcs / pkg or Catheter Edi, 6Fr, 50 cm, PHT free 5 pcs / pkg). Measurements will be performed using the esophageal transducer under two conditions: 2 hours in conventional ventilation (pressure controlled), 2 hours in NAVA ventilation and then again 2 hours in conventional ventilation (PC) for a total duration of 6 hours.The parameters of conventional ventilation will be left free at the choice of the neonatologist and will be identical between the two periods of conventional ventilation. The initial NAVA level will be defined by the neonatologist using pre-visualization curves. All signals will be recorded via an amplification and acquisition system. Values will be averaged over 100 cycles.

SUMMARY:
Congenital diaphragmatic hernia (CDH) is a congenital malformation associated with significant mortality and respiratory morbidity, particularly related to prolonged mechanical ventilation. NAVA (Neurally Adjusted Ventilatory Assist) is a recent technique that uses the recognition of the electrical activity of the patient's diaphragm (Edi) and delivers a synchronized proportional assisted ventilation. This technique has already been used in the newborn, especially premature and has shown many benefits. Only one study in the literature shows its feasibility in newborns with CDH. This technique seems interesting in the context of CDH because it would limit baro-trauma and improve synchronization. Before demonstrating the clinical benefits, it seems important to describe the effects on the respiratory physiology, in particular on work of breathing which can be estimated by the esophageal and trans-diaphragmatic pressure-time product obtained by an esophageal transducer. Our study is an innovative physiologic pilot study with the objective to describe work of breathing in neonates with CDH in post-surgical period in NAVA ventilation and in conventional ventilation using an esophageal transducer. It will provide the clinician with a physiological justification for the use of NAVA to rapidly improve the respiratory muscular dynamics of these patients. This study is a prerequisite for the realization of studies demonstrating the clinical benefit of NAVA ventilation on reduction of duration of ventilation and more generally on morbidity and mortality in the population of neonate with CDH.

ELIGIBILITY:
Inclusion Criteria:

* Neonate admitted to neonatal intensive care beyond 34 weeks of amenorrhea
* With a diagnosis of congenital diaphragmatic hernia having undergone a repair surgery.
* Necessary invasive ventilatory support by conventional ventilation
* Informed and signed consent of parents (and / or holders of parental authority)

Exclusion Criteria:

* Refusal of parents (and / or holders of parental authority) to participate in the study
* Contra-indication to the use of an oro or naso-gastric tube (oesophageal surgery)
* Child at risk of poor tolerance to the placement of the oesophageal pressure transducer (history of discomfort when placing a tube, weight <1500g)
* Central or neuromuscular neurological pathology which may affect respiratory control

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Work of breathing averaged over 100 consecutive cycles in NAVA ventilation and conventional ventilation | in post-surgical period during 6 hours
  Work of breathing is estimated by the esophageal and trans-diaphragmatic pressure-time product obtained by an esophageal transducer

SECONDARY OUTCOMES:
Patient-ventilator synchronization in NAVA | through study completion, an average of 1 year
  Comparison of the asynchrony indexes between the 2 modes (Number of asynchronies / Number of respiratory cycles)
Patient-ventilator synchronization in conventional ventilation | through study completion, an average of 1 year
  Comparison of the asynchrony indexes between the 2 modes (Number of asynchronies / Number of respiratory cycles)
Dynamic hyperinflation (intrinsic PEEP) in NAVA | through study completion, an average of 1 year
  Intrinsic PEEP average over 100 cycles
Dynamic hyperinflation (intrinsic PEEP) in conventional ventilation. | through study completion, an average of 1 year
  Intrinsic PEEP average over 100 cycles
Ventilation parameters: peak inspiratory pressure in NAVA | through study completion, an average of 1 year
  Evolution of the following parameters: peak inspiratory pressure, mean pressure, tidal volume, Ti / Ttot ration, FiO2
Ventilation parameters: mean pressure in NAVA | through study completion, an average of 1 year
  Evolution of the following parameters: peak inspiratory pressure, mean pressure, tidal volume, Ti / Ttot ration, FiO2
Ventilation parameters: tidal volume in NAVA | through study completion, an average of 1 year
  Evolution of the following parameters: peak inspiratory pressure, mean pressure, tidal volume, Ti / Ttot ration, FiO2
Ventilation parameters: Ti / Ttot ratio in NAVA | through study completion, an average of 1 year
  Evolution of the following parameters: peak inspiratory pressure, mean pressure, tidal volume, Ti / Ttot ration, FiO2
Ventilation parameters: FiO2 in NAVA | through study completion, an average of 1 year
  Evolution of the following parameters: peak inspiratory pressure, mean pressure, tidal volume, Ti / Ttot ration, FiO2
Ventilation parameters: peak inspiratory pressure in conventional ventilation | through study completion, an average of 1 year
  Evolution of the following parameters: peak inspiratory pressure, mean pressure, tidal volume, Ti / Ttot ration, FiO2
Ventilation parameters: mean pressure in conventional ventilation | through study completion, an average of 1 year
  Evolution of the following parameters: peak inspiratory pressure, mean pressure, tidal volume, Ti / Ttot ration, FiO2
Ventilation parameters: tidal volume in conventional ventilation | through study completion, an average of 1 year
  Evolution of the following parameters: peak inspiratory pressure, mean pressure, tidal volume, Ti / Ttot ration, FiO2
Ventilation parameters: Ti / Ttot ratio in conventional ventilation | through study completion, an average of 1 year
  Evolution of the following parameters: peak inspiratory pressure, mean pressure, tidal volume, Ti / Ttot ration, FiO2
Ventilation parameters: FiO2 in conventional ventilation | through study completion, an average of 1 year
  Evolution of the following parameters: peak inspiratory pressure, mean pressure, tidal volume, Ti / Ttot ration, FiO2
Physiological parameters indirectly evaluating work of breathing: esophageal swing in NAVA | through study completion, an average of 1 year
  Averages of the esophageal and diaphragmatic swings over 100 cycles in each period. Esophageal and diaphragmatic swings are physiological parameters obtained by the esophageal transducer which expressed muscle strength.
Physiological parameters indirectly evaluating work of breathing: diaphragmatic swing in NAVA | through study completion, an average of 1 year
  Averages of the esophageal and diaphragmatic swings over 100 cycles in each period. Esophageal and diaphragmatic swings are physiological parameters obtained by the esophageal transducer which expressed muscle strength.
Physiological parameters indirectly evaluating work of breathing: esophageal swing in conventional ventilation | through study completion, an average of 1 year
  Averages of the esophageal and diaphragmatic swings over 100 cycles in each period. Esophageal and diaphragmatic swings are physiological parameters obtained by the esophageal transducer which expressed muscle strength.
Physiological parameters indirectly evaluating work of breathing: diaphragmatic swing in conventional ventilation | through study completion, an average of 1 year
  Averages of the esophageal and diaphragmatic swings over 100 cycles in each period. Esophageal and diaphragmatic swings are physiological parameters obtained by the esophageal transducer which expressed muscle strength.
Clinical parameters of neonates: respiratory rate in NAVA | through study completion, an average of 1 year
  Evolution of clinical parameters (respiratory rate, heart rate, blood pressure) at the beginning and end of each period
Clinical parameters of neonates: heart rate in NAVA | through study completion, an average of 1 year
  Evolution of clinical parameters (respiratory rate, heart rate, blood pressure) at the beginning and end of each period
Clinical parameters of neonates: blood pressure in NAVA | through study completion, an average of 1 year
  Evolution of clinical parameters (respiratory rate, heart rate, blood pressure) at the beginning and end of each period
Clinical parameters of neonates: respiratory rate in conventional ventilation | through study completion, an average of 1 year
  Evolution of clinical parameters (respiratory rate, heart rate, blood pressure) at the beginning and end of each period
Clinical parameters of neonates: heart rate in conventional ventilation | through study completion, an average of 1 year
  Evolution of clinical parameters (respiratory rate, heart rate, blood pressure) at the beginning and end of each period
Clinical parameters of neonates: blood pressure in conventional ventilation | through study completion, an average of 1 year
  Evolution of clinical parameters (respiratory rate, heart rate, blood pressure) at the beginning and end of each period
Gas exchange: measurement of transcutaneous SaO2 in NAVA | through study completion, an average of 1 year
  Evolution of oxygenation parameters (SpO2) and transcutaneous CO2 (pCO2) during each period. SpO2 and pCO2 are measured continuously; average and median will be valued in each period of the study. No blood test will be required.
Gas exchange: measurement of transcutaneous pCO2 in NAVA | through study completion, an average of 1 year
  Evolution of oxygenation parameters (SpO2) and transcutaneous CO2 (pCO2) during each period. SpO2 and pCO2 are measured continuously; average and median will be valued in each period of the study. No blood test will be required.
Gas exchange: measurement of transcutaneous pCO2 in conventional ventilation | through study completion, an average of 1 year
  Evolution of oxygenation parameters (SpO2) and transcutaneous CO2 (pCO2) during each period. SpO2 and pCO2 are measured continuously; average and median will be valued in each period of the study. No blood test will be required.
Gas exchange: measurement of transcutaneous SaO2 in conventional ventilation | through study completion, an average of 1 year
  Evolution of oxygenation parameters (SpO2) and transcutaneous CO2 (pCO2) during each period. SpO2 and pCO2 are measured continuously; average and median will be valued in each period of the study. No blood test will be required.
Neonate comfort scores: COMFORT-BEHAVIOR score in NAVA | through study completion, an average of 1 year
  Evaluation of comfort (COMFORT-BEHAVIOR scale) at the beginning and at the end of each period.
Neonate comfort scores: COMFORT-BEHAVIOR score in conventional ventilation | through study completion, an average of 1 year
  Evaluation of comfort (COMFORT-BEHAVIOR scale) at the beginning and at the end of each period.

CONTACTS AND LOCATIONS:
Overall Officials: Lélia Dreyfus, MD, Principal Investigator — Service de Réanimation Néonatale- Hôpital Femme Mère Enfant- Hospices Civils de Lyon
Locations (1):
- Service de Réanimation Néonatale- Hôpital Femme Mère Enfant- Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dreyfus L, Butin M, Plaisant F, Claris O, Baudin F. Respiratory physiology during NAVA ventilation in neonates born with a congenital diaphragmatic hernia: The "NAVA-diaph" pilot study. Pediatr Pulmonol. 2023 May;58(5):1542-1550. doi: 10.1002/ppul.26357. Epub 2023 Mar 1. PMID 36807570